CLINICAL TRIAL: NCT06228209
Title: Tier - Palliative Care: A Population-based Care Delivery Model to Match Evolving Patient Needs to Palliative Care Services for Community-based Patients With Heart Failure or Cancer
Brief Title: Tier - Palliative Care For Patients With Advanced Heart Failure or Cancer
Acronym: TIER-PC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Laura Gelfman, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY-22-00591; 1R56NR020624-01 (NIH)
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Advanced Heart Failure; Advanced Non-colorectal Gastro-intestinal Cancer; Advanced Lung Cancer
Keywords: palliative care; community-based; advanced heart failure; advanced cancer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Before each research interview, subjects will be reminded not to tell the research coordinator to which study group they were assigned. In case of inadvertent unblinding of a blinded study team member, this team member will have to report the unblinding event to the PI. The study team member will not be allowed to collect data for the subjects whose group allocation they have inadvertently been unblinded to. A different, fully blinded study team member has to collect data for the respective subjects henceforth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tier - Palliative Care (Experimental): Patients/caregivers will be cared for by an interdisciplinary team that includes a social worker, nurse, community health worker, nurse practitioner, and physician.
  Interventions: Behavioral: Tier - Palliative Care
- Usual care (No Intervention): Patients will be cared for by the physician who treats their serious illness (cardiologist, oncologist, primary treating clinician) and other illnesses.

INTERVENTIONS:
Behavioral: Tier - Palliative Care — TIER-PC is an adaptive model of delivering palliative care that provides the right level of care to the right patients at the right time. It represents an adaption of the Mount Sinai PALLIATIVE CARE AT HOME (PC@H) program, which delivers home-based palliative care. TIER-PC increases the number and intensity of disciplines added to the patient's care team as their symptoms worsen and function declines.
  Arms: Tier - Palliative Care

SUMMARY:
TIER-PC is an adaptive model of delivering palliative care that provides the right level of care to the right patients at the right time. It represents an adaption of the Mount Sinai PALLIATIVE CARE AT HOME (PC@H) program, which delivers home-based palliative care. TIER-PC increases the number and intensity of disciplines added to the patient's care team as their symptoms worsen and function declines. In Tier 1, patients who are able to care for themselves and no/mild symptoms receive a community health worker (CHW) trained to elicit illness understanding in a culturally competent way. In Tier 2, for patients with poorer function and mild symptoms, a social worker (SW), trained in serious illness communication, joins the CHW to further elicit patients' goals and prognostic understanding while communicating symptom needs to their primary clinician. In Tier 3, as function decreases and symptoms increase, an advance practice nurse (APN) joins the CHW and SW to manage complex symptoms. Finally, in Tier 4, for those older adults with the poorest function and most complex symptoms, a physician joins the team to ensure that the most complex needs (e.g., end-of-life treatment preferences and multifaceted symptom control) are met. The CHW follows patients longitudinally across all tiers and re-allocates them to the appropriate tier based on their evolving needs.

DETAILED DESCRIPTION:
The study aims are:

* To evaluate the feasibility of enrolling patients into a study of TIER-PC; and
* To provide data on subject retention, randomization success, intervention fidelity and estimates of the efficacy of the TIER-PC intervention in improving patients' symptoms and quality of life, and reducing emergency department visits and hospitalizations.

This study will enroll 60 subjects with advanced non-colorectal gastrointestinal or lung cancer or advanced HF, 30 of which will be randomized to receive the study intervention and 30 of which will be randomized to receive usual care.

The expected study duration is 18 months from enrollment initiation to completion of data analysis consisting of a 52- week active enrollment period, a 3 month follow up period, and a three month data analysis period.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Heart Failure (HF) with two HF-related hospitalizations within the last 12 months or
* Advanced lung or non-colorectal gastrointestinal cancer (pancreatic, gastric, hepatobiliary, small bowel, esophageal) with one hospitalization within the last 6 months
* KPS > 50% (ECOG 0, 1 or 2)
* > 2 outpatient MSHS visits in prior 12 months
* Manhattan residence
* Capacity to provide informed consent
* English or Spanish fluency
* > 18 years of age

Exclusion Criteria:

* Diagnoses of both cancer and advanced HF
* Lung cancer with a driver mutation (e.g., EGFR) that confers a favorable prognosis and does not follow typical trajectory
* Patients with > 1 visit to Outpatient Supportive Oncology/Cardiology visit
* Patients with last visit to Outpatient Supportive Oncology/Cardiology < 3 months ago
* Previous receipt of a ventricular assist device or previous heart transplantation
* Receiving hospice care prior to study enrollment or enrolled in another study of a palliative care patient/caregiver intervention
* Living in a facility (subacute rehab, long-term care facility, hospice facility or residence)
* Callahan 6-Item Cognitive Screening score ≤3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-08-19 (Estimated); Study Completion 2026-08-19 (Estimated)

PRIMARY OUTCOMES:
The proportion of screened eligible patients | 3 months
  The proportion of screened eligible patients that are enrolled in the trial.

SECONDARY OUTCOMES:
The proportion of patients completing the final 3-month visit | 3 months
  The proportion of the patients completing the final 3-month visit among all enrolled patients.
Number of TIER-PC intervention visits received per patient per month | 3 months
  The fidelity to intervention is defined as the number of TIER-PC intervention visits received per patient per month in the TIER-PC arm during the follow-up period.
Edmonton Symptom Assessment Scale (ESAS) | 3 months
  Patient symptoms will be measured (e.g., pain, shortness of breath) using the 9-item Edmonton Symptom Assessment Scale (ESAS) validated for serious illness. Each item is 10-point scale, total score ranges 0 (no symptoms) - 90 (worst severity), with higher scores indicating worse symptom severity.
Quality of Life measured using Functional Assessment of Chronic Illness Therapy-Palliative Care Scale (FACIT-Pal) | 3 months
  Quality of life (QoL) using the Functional Assessment of Chronic Illness Therapy-Palliative Care Scale (FACIT-Pal), a 46-item QoL questionnaire validated in patients with advanced disease. Each item is scored on a 5-point Likert scale from 0 (not at all) - 4 (very much). Total score ranges 0-184, with higher scores indicating better quality of life.
Number of participant emergency department (ED) visits | 3 months
  Number of participant ED visits
Number of participant hospitalizations | 3 months
  Number of participant hospitalizations
Number of participant hospital days | 3 months
  Number of participant hospital days
Patient-Reported Goals of Care Discussion (GOCD) | 3 months
  Patient report of goals of care discussions. Single item on GOCD with clinician. Response: Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Laura P Gelfman, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  For individual participant data meta-analysis. Proposals should be directed to Arushi.Arora@mssm.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website, to be determined.